CLINICAL TRIAL: NCT06644274
Title: The Value of 68Ga-grazytracer PET in Monitoring Responses to Immunotherapy of Gastrointestinal Malignancies
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-278
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Gastrointestinal Malignancies
Keywords: 68Ga-grazytracer PET/CT; gastrointestinal malignancies; Immunotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosis of gastrointestinal malignancies: Patients diagnosis of gastrointestinal malignancies require immunotherapy or combination immunotherapy after evaluation according to clinical guidelines

SUMMARY:
This study aims to investigate the value of 68Ga-grazytracer in predicting the efficacy of immunotherapy for gastrointestinal malignancies.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-grazytracer PET/CT after 3 cycles of immunotherapy to evaluate response. The imaging response measurements will be compared with the histopathological or clinical assessment results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and clinical diagnosis of gastrointestinal malignancies requiring immunotherapy or combination immunotherapy after evaluation according to clinical guidelines.
2. Signed and dated informed consent form.
3. Commitment to comply with research procedures and co-operation in the implementation of the full research process.
4. The patient is in good general condition with an expected survival of > 6 months.
5. aged 18-75 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction.
3. Pregnant women and women who may be pregnant, women who are breastfeeding.
4. Non-compliant person.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the responses to immunotherapy of gastrointestinal malignancies | up to about 10 weeks
  The value of 68Ga-grazytracer PET in monitoring responses to immunotherapy of gastrointestinal malignancies
Standardized uptake value(SUV) | up to about 10 weeks
  SUV of 68Ga-grazytracer uptake on PET/CT images for tumor lesions
Target-to-background ratio(TBR) | up to about 10 weeks
  68Ga-grazytracer uptake ratio of tumor lesions to mediastinum and liver blood pool on PET/CT images.

SECONDARY OUTCOMES:
Progress free survival | 1 years
  Progress free survival
Overall survival | 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No